CLINICAL TRIAL: NCT02208804
Title: Surefire Infusion System vs. Standard Microcatheter Use During Holmium-166 Radioembolization for the Treatment of Colorectal Liver Metastases (SIM Trial)
Brief Title: Surefire Infusion System vs. Standard Microcatheter Use During Holmium-166 Radioembolization
Acronym: SIM
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Maurice A.A.J. van den Bosch, Prof. dr., UMC Utrecht
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 14-287/D
Record Dates: First submitted 2014-07-31; First posted 2014-08-05 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Colorectal Neoplasms; Neoplasm Metastasis; Liver Diseases; Digestive System Neoplasms
Keywords: Colorectal Cancer Liver Metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Liver Diseases; Digestive System Neoplasms | interventions — Microspheres

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surefire Infusion System (Experimental): Hepatic arterial administrations using the Surefire Infusion System
  Interventions: Device: Holmium-166-poly (L-lactic acid) microspheres
- Standard End-hole Microcatheter (Active Comparator): Hepatic arterial administrations using the standard end-hole microcatheter
  Interventions: Device: Holmium-166-poly (L-lactic acid) microspheres

INTERVENTIONS:
Device: Holmium-166-poly (L-lactic acid) microspheres

SUMMARY:
The objective of the SIM trial is to investigate whether using the Surefire Infusion System during holmium-166 radioembolization increases the posttreatment tumor to non-tumor activity concentration ratio, compared with using a standard end-hole microcatheter.

DETAILED DESCRIPTION:
Study design: clinical within-subject randomized controlled trial.

Study population: 25 patients with unresectable, chemorefractory, liver-dominant colorectal liver metastases.

Intervention: scout and therapeutic doses of holmium-166 microspheres will be administered in the left and right hepatic artery during two sequential angiography procedures on the same day. In all subjects, the use of the Surefire Infusion System and the standard end-hole catheter will be randomly allocated to the infusion site (left and right hepatic artery).

Baseline and follow-up investigation: at baseline and during follow-up, patients will undergo physical examination and laboratory investigations for toxicity assessment, and a whole-body 18F-FDG-PET + dual-phase liver CT (at baseline and 3-months follow-up) for tumor response assessment. After the scout procedure and therapeutic procedure, a holmium-166 SPECT/CT will be obtained for the assessment of the microsphere distribution.

Main study parameters/endpoints:

The primary endpoint is the tumor to non-tumor activity concentration ratio on SPECT/CT.

Secondary endpoints include mean absorbed doses of radioactivity in tumorous and healthy liver tissue, tumor response, the predictive value of holmium-166 scout dose and infusion efficiency. These endpoints will be compared between the Surefire Infusion System and standard microcatheter infusions. A dose-response relationship, clinical toxicity and overall survival will be assessed for the entire cohort.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Histopathologically confirmed diagnosis of adenocarcinoma of the colon or rectum
* Hepatic metastases with measurable morphological appearance (≥ 1 cm) on cross sectional imaging, located in the right and left hepatic arterial perfusion territory
* Unresectable, liver dominant disease
* Progressive disease after second line chemotherapy or no further chemotherapeutical treatment options due to severe side effects or unwillingness of the patient to undergo systemic chemotherapy
* Age ≥ 18 years
* Expected adequacy of follow-up

Exclusion Criteria:

* World health organization performance score > 2
* Inadequate bone marrow function (hemoglobin < 6.0 mmol/l, leukocyte count < 3.0 x 109/l, platelet count < 75x 109/l), inadequate liver function (bilirubin > 35 µmol/l, aspartate aminotransferase / alanine aminotransferase (AST/ALT) > 5 x upper limit of normal (ULN)) or inadequate renal function (creatinine > 1.5 x ULN)
* Prior hemihepatectomy
* Compromised biliary system (biliary stent or hepaticojejunostomy)
* Child Pugh score B7 or worse
* Active hepatitis B or C
* Main portal vein thrombosis on CT (or previous portal vein embolization)
* Severe celiac axis stenosis on CT
* Unsuitable hepatic arterial anatomy on CT
* Treatment with systemic chemotherapy within 4 weeks prior to radioembolization
* Previous participation in a study classified as class III by a radiation safety committee
* Bleeding diathesis
* Pregnancy or breast feeding
* Life expectancy < 3 months
* Patients who are declared incompetent
* Any condition that prevents from safe treatment with radioembolization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Posttreatment tumor to non-tumor activity concentration ratio on SPECT/CT | 5 days after treatment

SECONDARY OUTCOMES:
Mean absorbed radiation doses in tumorous and healthy liver tissue on SPECT/CT | 5 days after treatment
Posttreatment tumor response on CT and 18F-FDG-PET | 3 months after treatment
Predictive value of the holmium-166 scout dose | On the day of treatment
Dose-response relationship between tumor absorbed doses on SPECT/CT and tumor response on CT and 18F-FDG-PET | 3 months after treatment
Infusion efficiency | On the day of treatment
  Defined as the percentage of calculated treatment activity that was administered
Overall survival | From date of treatment until the date of death from any cause, assessed up to 1 year
Clinical and laboratory toxicity | Up to 3 months after treatment
  According to Common Terminology Criteria for Adverse Events version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Maurice AAJ van den Bosch, Prof. dr., Principal Investigator — UMCU Utrecht, The Netherlands; Max A Viergever, Prof. dr. ir., Study Director — UMC Utrecht, The Netherlands
Locations (1):
- Department of Radiology and Nuclear Medicine, University Medical Center Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] van Roekel C, van den Hoven AF, Bastiaannet R, Bruijnen RCG, Braat AJAT, de Keizer B, Lam MGEH, Smits MLJ. Use of an anti-reflux catheter to improve tumor targeting for holmium-166 radioembolization-a prospective, within-patient randomized study. Eur J Nucl Med Mol Imaging. 2021 May;48(5):1658-1668. doi: 10.1007/s00259-020-05079-0. Epub 2020 Oct 31. PMID 33128132
- [Derived] van den Hoven AF, Prince JF, Bruijnen RC, Verkooijen HM, Krijger GC, Lam MG, van den Bosch MA. Surefire infusion system versus standard microcatheter use during holmium-166 radioembolization: study protocol for a randomized controlled trial. Trials. 2016 Oct 25;17(1):520. doi: 10.1186/s13063-016-1643-3. PMID 27782851